CLINICAL TRIAL: NCT01988402
Title: Does Allopurinol Prolong a Treated, Acute Gout Flare?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jay B. Higgs, MD, Program Director, Rheumatology Fellowship, 59th Medical Wing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWH20070235H
Record Dates: First submitted 2013-11-06; First posted 2013-11-20 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Gout
Keywords: gout; allopurinol
MeSH Terms: conditions — Gout | interventions — Allopurinol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Active Comparator): Patients in this arm receive allopurinol, 100 mg daily for 14 days and then 200 mg daily for 14 days
  Interventions: Drug: allopurinol
- Sugar pill (Placebo) (Placebo Comparator): Patients in this arm receive one placebo (sugar) pill per day for 14 days then 2 placebo pills for 14 days.
  Interventions: Drug: Placebo (sugar pill)

INTERVENTIONS:
Drug: allopurinol
  Arms: Allopurinol
Drug: Placebo (sugar pill)
  Arms: Sugar pill (Placebo)

SUMMARY:
This is a double blind placebo controlled study to determine whether starting allopurinol during a treated acute gout attack will have any effect on the duration of the attack.

DETAILED DESCRIPTION:
Traditional teaching holds that starting allopurinol during an acute gout attack will prolong the attack. Recent expert opinion from the American College of Rheumatology Guidelines is that allopurinol may be started during an acute, treated gout attack. This study is designed to test the hypothesis that allopurinol does not prolong an acute, treated gout attack. Patients will either take allopurinol capsules or and identical capsule containing no allopurinol (placebo) over 28 days, starting within 72 hours of a gout attack that is being treated with other standard measures. During the study, neither the patient nor the examiner will know what pills are being taken. The time to resolution of the attack is the primary outcome measure. Pain level, serum uric acid level, and complications of therapy will also be monitored. A minimum of 32 patients completing the study are needed for a meaningful conclusion.

ELIGIBILITY:
Inclusion Criteria requires both of:

* Crystal proven gout, and
* An acute gout attack within 72 hours of first treatment

Plus one of the following:

* At least 2 gout attacks in past 12 months
* Tophus
* Nephrolithiasis
* 24hr urine uric acid greater than 1000mg

Exclusion Criteria:

* Inability to return for examinations
* Glomerular filtration rate (calculated) less than 50 milliliters per minute
* Allopurinol use in past 6 months
* Ongoing cancer therapy
* Concomitant azathioprine or cyclophosphamide
* Any one of the following liver enzymes greater than 1.25 times the upper limit of normal:

  * AST [Aspartate aminotransferase]
  * ALT [Alanine aminotransferase]
  * alkaline phosphatase
* Pre-gout pain in involved joint of more than 3 on a scale of 1-10
* Neurologic deficit around the involved joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay B Higgs, MD, Principal Investigator — 59th Medical Wing
Locations (1):
- Wilford Hall Ambulatory Surgical Center, Lackland Air Force Base, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 patients were enrolled which achieved a completer number of 31. This was one short of the original completer target of 32. Power analysis suggested that a much larger number would have been required to achieve statistical power, and that enrolling 1-2 more subjects would not have contributed to the data.
Groups:
- Allopurinol: Patients in this arm receive allopurinol, 100 mg daily for 14 days and then 200 mg daily for 14 days
  allopurinol
- Sugar Pill (Placebo): Patients in this arm receive one placebo (sugar) pill per day for 14 days then 2 placebo pills for 14 days.
  Placebo (sugar pill)
Period: Overall Study
Arm/Group | Allopurinol | Sugar Pill (Placebo)
Started | 16 | 19
Completed | 14 | 17
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allopurinol | Sugar Pill (Placebo) | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Mean (Full Range); unit: Years] | 61 [40 to 84] | 53 [31 to 68] | 57 [31 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 14 | 19 | 33
Disease duration [Mean (Full Range); unit: years] | 5.5 [0 to 20] | 4.9 [0 to 17] | 5.2 [0 to 20]
number of prior attacks [Mean (Full Range); unit: number] | 3.7 [0 to 12] | 6.58 [1 to 35] | 5.2 [0 to 35]
participants with history of nephrolithiasis [Number; unit: participants] | 4 | 1 | 5
participants with tophi [Number; unit: participants] | 6 | 6 | 12
Participants with erosions [Number; unit: participants] | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Resolution of the Acute Gout Attack
Description: The primary outcome unit of measurement is time (in days) to resolution of the acute gout attack
Time Frame: 1-28 Days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Allopurinol | Sugar Pill (Placebo)
Number analyzed (Participants) | 14 | 17
days | 15.4 (7.9) | 13.4 (7.8)
Statistical Analysis 1: Comparison: Allopurinol vs Sugar Pill (Placebo); Test type: Superiority or Other; p = 0.5, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Day 28
Description: Patient rated pain on a Likert pain score of 0-10
Time Frame: Pateints are assessed at five time intervals over 28 days: days 1, 3-4, 10-15, 20-25, and 28; Day 28 reported
Measure: Mean (95% Confidence Interval); unit: units on a Likert scale
Arm/Group | Allopurinol | Sugar Pill (Placebo)
Number analyzed (Participants) | 16 | 19
units on a Likert scale | 1.79 [0 to 4] | 2.0 [0 to 4]

3. Secondary Outcome: Physician Global Assessment of Gout Activity at Day 28
Description: Physician rated gout activity is measured on a Likert scale 0-10.
Time Frame: Pateints are assessed at five time intervals over 28 days: days 1, 3-4, 10-15, 20-25, and 28; Day 28 reported
Measure: Mean (95% Confidence Interval); unit: units on a Likert scale
Arm/Group | Allopurinol | Sugar Pill (Placebo)
Number analyzed (Participants) | 16 | 19
units on a Likert scale | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Serum Uric Acid Level
Description: Blood test (serum) for uric acid level
Time Frame: day 28
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Allopurinol | Sugar Pill (Placebo)
Number analyzed (Participants) | 14 | 17
mg/dl | 6.4 (1.0) | 8.2 (1.0)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Allopurinol | Sugar Pill (Placebo)
Serious Adverse Events (participants affected / at risk) | 1/16 | 2/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopurinol (N=16) | Sugar Pill (Placebo) (N=19)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
elevated liver enzymes (Gastrointestinal disorders) | 0 | 1
nausea and vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes